CLINICAL TRIAL: NCT05139407
Title: Effect of Six Weeks Content Knowledge Workshop on Written Test Performance Among Physical Education Students in China
Brief Title: Experimental Intervention on the Influence of Six Weeks' Content Knowledge on Students' Written Test Achievement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Yongqi Gao, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Yongqi Gao
Record Dates: First submitted 2021-08-28; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Educational Problems; Student Burnout
Keywords: Content knowledge; Written test perfofmance; Students
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Individual trials cannot be made public before publication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshop (Experimental): The workshop is to discuss methods in various fields through activities, discussions, and lectures. It is an academic way to encourage participation, innovation, and predict solutions, suitable for people from different positions and ethnic groups to think, discuss, and communicate.
  Each Intervention includes information relevant to how the Intervention was administered to participants in the associated Arm.
  Workshop intervention for students: basketball training plan, basketball lesson plan, energy supply in muscle exercise, exercise prescription, track, and field mapping, basketball rules. All patients were intervened according to the frequency of 3 hours/once a week.
  Interventions: Diagnostic Test: Teaching intervention
- Oral examination (Experimental): The oral examination is a way of examination, which requires the examination to answer questions orally. Content intervention includes the comment, teacher's question and answer, proposition explanation, and proposition debate. In addition, each Intervention provides information relevant to how the Intervention was administered to students in the associated Arm.
  Specific interventions for students: basketball training plan, basketball lesson plan, energy supply system, exercise prescription formulation, track and field venue planning, basketball game rules. All oral examinations take 90 minutes/once/week.
  Interventions: Diagnostic Test: Teaching intervention

INTERVENTIONS:
Diagnostic Test: Teaching intervention — Different teaching methods are used to teach the experimental group and the control array in the classroom.

SUMMARY:
Brief Summary .

This experiment aims to use two different teaching methods to intervene in students' learning and find out which teaching method is more conducive to improving students' written test achievement. The experiment will use a 6-the investigator seek workshop intervention to enhance students' written test achievement. The investigation is divided into workshop groups and standard teaching groups. The most significant difference better investigators the two groups are that the workshop group has oral links and guarantees. The similarities between investigators in the two groups are teacher qualifications, intervention time, content, and research objects.

Based on content knowledge learning, content knowledge is divided into six categories for detailed intervention. First, the investigators will do a 6-the investigator seek intervention for two groups (workshop style and standard teaching style). The difference better investigators two is whether there is a video teaching link, and the same is that there are oral links. The entire experiment was carried out in the classroom with the school's consent. Use written exams to check student scores. Students have special teachers responsible for teaching specific content knowledge during class, standard learning after class does not require special care, and the experiment is not risky.

Hypothesis including as follow:1 ) General Hypothesis. There is no significant difference in the written test results of the prior theoretical knowledge 、health promotion knowledge、 physical exercise knowledge control group, with experimental group performance among PE students in China. 2) Specific Hypothesis. The specific hypothesis of this study is to investigate the effect of a 6-weeks content knowledge workshop on written test performance among PE students in China. The detailed hypothesis is: There is no significant difference between the control and experimental groups in the sports training design、the teaching design 、the muscle function system、the exercise physiology、the competition venue planning、the referee rules written test performance among PE students in China.

DETAILED DESCRIPTION:
Detailed Description

Location.The University of China. In terms of students, the proportion of people who choose to work is high, while the proportion of people who choose to continue their postgraduate entrance tests is negligible. Sports graduates account for 70% of a Province, and students have not participated in workshop study. On the school side, the school has perfect teaching equipment to meet the experimental requirements, conducive to better completion.

The analysis of intervention Plan-same characteristics mainly includes two parts: Teacher qualification and student qualifications. In the first part, workshop group and standard teaching group, teacher Qualification, same qualification and titles, both have one same teacher majors: physical education, similar experience: minimum more than ten years.No students have received this courses before the study. The second part is the age, major and educational background of students. For example, students with similar educational backgrounds, aged 19 and 25, are all majors in physical education.No students have received these courses before the study.

This part discusses the details of the 6-the investigator seeks workshop and standard teaching intervention. First and foremost, CK includes three categories. Then, the deeper level is divided into six parts: methods and plans, class hour teaching plan, muscle exercise, energy supply, breathing and exercise circulation and exercise, athletic and basketball venue, basketball, and football rules. On the other hand, there are two lessons; each class is 1.5 hours.

This is a one-class training plan, mainly divided into other structures. A training session explicitly includes three parts.

To start with, the intervention content includes step 1-An, an overview, and introduction, step 2-Students formed groups, step 3-Oral test assessment. The first part includes: The teacher introduced the purpose of the study, expectations, and discussion of the principles of sports training design. Next, the investigators learn to design, muscle function, and exercise physiology system-rest time.

The second part includes introducing the purpose of the study, expectations, and discussion of the principles of sports training design. They the investigators learn content related to design and muscle function and exercise physiology systems. Rest time Divided into three groups and rotated roles of teacher, students, 8 / group. They the investigators learn by the reciprocal peer learning instructional model.

The third part includes introducing the purpose of the study, expectations, and discussion of the principles of sports training design. They the investigators learn content related to design and muscle function and exercise physiology systems. Rest time Divided into three groups and rotated roles of teacher, students, 8 / group. They the investigators learn by the reciprocal peer learning instructional model. Students the investigators prompted to switch teacher roles, student every 10 min-evaluation through check sheets and oral test ( 90% or better correct and the investigators ).

ELIGIBILITY:
1. Inclusion Criteria:

   1. Students whose age meets the requirements.
   2. Students majoring in physical education in Ningxia University.
   3. Students who voluntarily participate and pass the qualification assessment.
   4. Students who can complete the experimental intervention plan.
   5. Students who have not participated in the examination and training.
2. Exclusion Criteria:

   1. Excluded because age of not meeting inclusion criteria
   2. Drop out be absent with leave、refuse to participate;
   3. Students who are often absent from school and late.
   4. Students who have already taken the exam.
   5. Not a college student in Ningxia University.

Ages: 21 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Random, unlimited
Enrollment: 26 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Students' written test achievements | 1 week -7 weeks
  Primary outcome measure information: students' content knowledge, the higher the students' written test achievement, the more significant the intervention.
  Title: Name of the specific primary outcome measure-written test. Description: Overview of Six parts content measurement. i.Measurement before Ist week and Measurement after the sixth week ii. Overall sample was written test achievements written test is 100, and the time of each test is 2 hours.
  Time Frame,1-6 weeks, Used in the written test achievement Calculation for each primary outcome measure Including one basketball lesson training plan in the first week, one basketball lesson plan in the second week, Energy supply in muscle exercise in the third week, Exercise prescription in the fourth week, The fifth week of Track and field venue planning and the sixth week of Track Meet rules. Each content knowledge measurement includes oral examination performance must be over 95, and each measurement time is 90 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: YONGQI GAO, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- China, Ningxia ,Ningxia University, Yingchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No
This research belongs to the need of personal doctoral thesis experiment and cannot be shared before publication.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23204206/

DOCUMENTS (1):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT05139407/Prot_000.pdf